CLINICAL TRIAL: NCT00870272
Title: A Randomized Study of Sublingual and Buccal Misoprostol Administration Following Mifepristone 200 mg for Abortion up to 63 Days Gestation
Brief Title: Study of 400mcg Sublingual Versus 400mcg Buccal Misoprostol Following 200mg Mifepristone for Medical Abortion up to 63 Days Last Menstrual Period (LMP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Beverly Winikoff/President, Gynuity Health Projects
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.2.0
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Abortion, Induced
Keywords: Medical Abortion; Mifepristone; Misoprostol; Sublingual administration; Buccal administration
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 400mcg sublingual misoprostol
  Interventions: Drug: Misoprostol
- 2 (Active Comparator): 400mcg buccal misoprostol
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 400mcg misoprostol taken sublingually or buccally

SUMMARY:
This open-label, randomized study is being conducted to determine whether a dose of 400 mcg of buccal misoprostol (i.e., in the cheek) taken 24 hours following administration of mifepristone 200 mg is as effective and acceptable at inducing an abortion compared with misoprostol taken sublingually (under the tongue). Women presenting for voluntary termination of intrauterine pregnancy with gestational ages of <63 days will be offered the option of participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than or equal to 63 days
* General good health including absence of conditions which contraindicate the use of mifepristone and misoprostol for pregnancy termination; and
* Willing to provide an address and/or telephone number for purposes of follow-up.

Exclusion Criteria:

* Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass
* IUD in place
* Chronic renal failure
* Concurrent long-term corticosteroid therapy
* History of allergy to mifepristone, misoprostol or other prostaglandin
* Hemorrhagic disorders or concurrent anticoagulant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Comparison of safety and efficacy of 2 different routes of misoprostol after mifepristone administration | July 2007-March 2009

SECONDARY OUTCOMES:
Side effects experienced | July 2007- March 2009

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Sheila Raghavan, MSc, Study Director — Gynuity Health Projects
Locations (1):
- State University of Medicine and Pharmacy, Chisinau, Moldova